CLINICAL TRIAL: NCT00274326
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind Trial Evaluating the Effect of a Vasopressin V2 Receptor Antagonist (SR121463B) on Serum Sodium in Patients With Dilutional Hyponatremia
Brief Title: DILIPO (DILutIonal HyPOnatremia)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5816
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2008-09-15 (Estimated); Status verified 2008-09

CONDITIONS: Congestive Heart Failure
Keywords: Hyponatremia
MeSH Terms: conditions — Heart Failure; Hyponatremia | interventions — satavaptan

INTERVENTIONS:
Drug: SR121463B

SUMMARY:
Primary:

* To assess the efficacy of SR121463B in correcting hyponatremia in patients with dilutional hyponatremia other than SIADH or cirrhosis

Secondary:

* To assess the long-term efficacy of SR121463B in maintaining normonatremia in these patients
* To assess the safety and tolerability of SR121463B

DETAILED DESCRIPTION:
SR121463B is an orally effective non-peptide, potent, and highly selective V2 receptor antagonist causing free water elimination in animals and humans

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients aged 18 higher
* Dilutional Hyponatremia with serum sodium between 115 and 132 mmol/L
* Ability to give written informed consent (the informed consent may be signed by a legally authorized representative if the patient is unable to sign)

Exclusion Criteria:

* Presence of known or untreated adrenal insufficiency, SIADH or cirrhosis, or hyperthyroidism
* Presence of signs of hypovolemia
* Administration of other V2 receptor antagonists or demeclocycline or lithium within one month and urea within two days prior to study drug administration
* Presence of uncontrolled diabetes with fasting glycemia ³ 200 mg/dL (³ 11.09 mmol/L)
* Patients considered by the Investigator unsuitable candidates to receive an investigational drug (e.g., presence of any neurological symptoms that may worsen in five days, based on the judgment of the Investigator, or presence of any neurological symptoms for which the persistence of hyponatremia over several days may be deleterious)
* Administration of inducers of CYP3A4 (phenobarbital, phenytoin, rifampin, Saint John's Wort) or potent and moderate inhibitors of CYP3A4 within two weeks prior to study drug administration
* Presence or history of allergic reaction to SR121463B8
* Previous study with SR121463B
* Inadequate hematological, renal, and hepatic functions: hemoglobin (Hb) < 9 g/dL, neutrophils < 1,500/mm3, platelets < 100,000/mm3, serum creatinine > 175 mol/L (or clearance of creatinine < 30 mL/min for sites where Ethics Committees require this parameter), serum alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 2 x upper limit of normal (ULN)
* QTCB 500 ³ ms
* Positive pregnancy test and absence of medically approved contraceptive methods (e.g., surgical sterilization of more than one month duration, oral contraception or intrauterine device in combination with either diaphragm, condom, or spermicide) for females of childbearing potential
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2005-05; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
EFFICACY:Serum Sodium
SAFETY:Physical examination, vital signs, adverse events, electrocardiogram, hematology, serum chemistry
PHARMACOKINETICS:Plasma SR121463B concentrations

SECONDARY OUTCOMES:
Weight; EQ-5D and pharmaco-economic assessments

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ter-Minassian, MD, Study Chair — Sanofi
Locations (15):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- sanofi-aventis Australia & New Zealand administrative office, Macquarie Park, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Bromma, Sweden

REFERENCES:
- [Derived] Aronson D, Verbalis JG, Mueller M, Krum H; DILIPO investigators. Short- and long-term treatment of dilutional hyponatraemia with satavaptan, a selective arginine vasopressin V2-receptor antagonist: the DILIPO study. Eur J Heart Fail. 2011 Mar;13(3):327-36. doi: 10.1093/eurjhf/hfq226. Epub 2011 Jan 3. PMID 21199833
- See also: Related Info — http://www.sanofi-aventis.com